CLINICAL TRIAL: NCT02716051
Title: Initial Staging of Bronchopulmonary Neoplasia: Whole-body MRI Versus Pet Scanner
Brief Title: Wholebody MRI In Lung Cancer StagiNg
Acronym: WISLON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: I15037/WILSON
Record Dates: First submitted 2016-03-14; First posted 2016-03-23 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRI (Experimental): Wholebody MRI with cardio-pulmonary synchronization At day 1 , at the afternoon, patient will undergo an MRI analysis.
  Interventions: Device: MRI
- PET (Active Comparator): At day 1 , in the morning, patient will undergo an PET analysis
  Interventions: Device: PET

INTERVENTIONS:
Device: MRI — Whole body MRI with cardiac and pulmonary synchronization
  Arms: MRI
Device: PET
  Arms: PET

SUMMARY:
Magnetic Resonnace Imaging (MRI) and Positron Emission Tomography (PET) can be both used in detection of nodes in patients with cell lung cancer (NSCLC).

However, the cardiorespiratory synchronization in the MRI, allowing acquisition of synchronous images with breathing and heart movements should increase the sensitivity of detection of pathologic mediastinal lymph nodes.

Given its high sensitivity, whole-body MRI with diffusion could possibly be at least as informative as PET, while being less expensive, not radiant.

The purpose of this study is to evaluate the performance of whole-body MRI with diffusion with cardiorespiratory synchronization, on the detection of mediastinal nodes (which are known to be less well detected by MRI) compared to PET.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years,
* Neoplasia bronchopulmonary (SCLC and NSCLC) newly diagnosed,
* Patient potentially eligible for curative treatment, but no no treatment started,
* Patients for whom a PET scan and MRI are planned

Non Inclusion Criteria:

* claustrophobia,
* Implantable Medical Device
* not compatible pacemaker type or heart valve, metal splinters eye)
* Pregnant or lactating women,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Th consistency of the locations of mediastinal lesions | Day 1
  Node localization according to MRI and PET scan measurements on the same day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No